CLINICAL TRIAL: NCT04397328
Title: Safety and Efficacy of Post-exposure Prophylaxis With Hydroxychloroquine (HCQ) for the Prevention of COVID-19 in High-risk Older Individuals in Long-term and Specialized Care: A Double-blind Randomized Control Trial
Brief Title: COVID-19 PEP- High-risk Individuals in Long-term and Specialized Care - Canada
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study Withdrawn
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 9881
Record Dates: First submitted 2020-05-13; First posted 2020-05-21 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2020-05

CONDITIONS: COVID-19
Keywords: COVID-19; Hydroxychloroquine; Double Blind Randomized Control Trial; Prophylaxis; High risk; Long term / specialized care
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydroxychloroquine 200mg (Experimental): Regular Dose 400mg orally once, followed in 8 hours by 400mg, then 200mg twice a day for 4 consecutive days (5 days in total) Modified Dose 400mg orally once, followed in 8 hours by 400mg, then 200mg once a day for 4 consecutive days (5 days in total) Modified doses are for individuals with body weight below 40 kg, renal impairment with a creatinine clearance less than 10mls/min or QTc interval greater than 480 but less than 500.
  Interventions: Drug: Hydroxychloroquine
- Placebo Arm (Placebo Comparator): The placebo arm will be matched to study drug to maintain the study blind. Regular Dose Placebo 2 tabs once, followed in 8 hours by 2 tabs, then 1 tab twice a day for 4 consecutive days (5 days in total) Modified Dose Placebo 2 tabs once, followed in 8 hours by 2 tabs, then 1 tab once a day for 4 consecutive days (5 days in total) Modified doses are for individuals with body weight below 40 kg, renal impairment with a creatinine clearance less than 10mls/min or QTc interval greater than 480 but less than 500.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine vs placebo (1:1 design) double blind intervention
  Arms: Hydroxychloroquine 200mg
Drug: Placebo — Hydroxychloroquine vs placebo (1:1 design) double blind intervention
  Arms: Placebo Arm

SUMMARY:
Older adults are at the highest risk of complications and severe illness for 2019-nCoV infections. Hydroxychloroquine (HCQ), an emerging chemoprophylaxis, which holds clinical and mechanistic plausibility, will help to reduce disease incidence and mitigate disease severity across in-patient settings. This study is designed to assess the safety and efficacy of post-exposure prophylaxis with hydroxychloroquine (HCQ) for the prevention of Coronavirus Infectious Disease-19 (COVID-19) in high-risk older individuals in long-term and specialized care.

DETAILED DESCRIPTION:
Rationale: HCQ blocks SARS-CoV-2 entry into host cells in vitro, and it also has immunomodulatory effects; therefore, it may be effective in reducing viral presence and inhibiting immunopathological mechanisms of COVID-19 in patients if administered before manifestation of clinical symptoms.

Hypothesis: the investigators hypothesize that prophylactic HCQ treatment in high-risk individuals Long Term Care (LTC) and Specialized Care (SC) settings post confirmed exposure to SARS-CoV-2 will reduce morbidity and mortality to COVID-19 via a) reduced viral presence during the acute phase of the infection, and b) inducing protective immune cell populations, c) reducing the production of inflammatory cytokines in peripheral blood.

Objectives:

Test if HCQ can prevent the development of COVID-19 in high-risk individuals in institutions which provide LTC or SC after known accidental exposure to the SARS-CoV-2.

Test if early presumptive therapy in asymptomatic high-risk individuals exposed to SARS-CoV-2 can limit disease progression and acute care hospitalization.

Study drug or placebo initiated after exposure, but before symptoms of elevated temperature, cough, or shortness of breath.

If the exposed patients developed respiratory symptoms, specifically fever, cough or dyspnea, the blinded treatment will be continued and usual supportive care added as per clinician preference. If antiviral or immunomodulatory therapy is recommended, the patient treatment allocation will be unblinded, and treatment may be administered as per clinician preference with consideration of locally available agents.

Safety will be closely monitored during the study conduct with safety labs and 6 lead ECGs at baseline, day 2, 5, 12, and 19

ELIGIBILITY:
Inclusion Criteria:

1. Age over 40 with two or more high-risk comorbidities that have been found to confer a higher risk of mortality including but not limited to :

   chronic lung disease to include: Chronic obstructive lung disease, interstitial lung disease or diffuse parenchymal disease moderate to severe asthma
   * Cardiac conditions to include: recent myocardial infarction (within the last three months) or poorly controlled heart failure
   * severe obesity (body mass index [BMI] of 40 or higher)
   * Diabetes (type 1 or 2)
   * chronic kidney disease undergoing dialysis
   * liver cirrhosis

   OR Age over 60.
2. Patient/resident in an Institute (to include a rehabilitation, long term care facility, mental health facility or veteran's care) that provides bed-based care in shared semi-private or ward rooms (i.e. two or more to a room) with a patient with confirmed COVID-19 for at least 6 hours in the absence of contact and droplet precautions.
3. Exposure with a documented or suspected COVID-19 case or from a symptomatic ( defined as common symptoms of COVID-19 including but not limited to fever, lethargy, dry cough, shortness of breath) health care worker providing direct patient contact within 3 feet without a mask for > 15min or any physical contact with the staff. Exposure may occur in single or shared bedrooms. Exposure may occur in a common dining or activity or sitting area. Any patient sharing a room or within 3 feet for > 15min or any physical contact without a mask will be considered as a contact. Patients or staff are considered as infectious for 48hrs before any symptoms onset and until masked or cleared by 2 negative swabs.
4. No prior treatment with acetaminophen or NSAIDs or willing to stop present prescription of regular or PRN acetaminophen.
5. Informed consent (in person or by telephone/e-mail with SDM)

Exclusion Criteria:

1. Greater than 96 hours since last exposure
2. Presence of fever (T>37.8), new onset cough, or shortness of breath at enrollment
3. A baseline O2 saturation less than 90% (as measured by pulse oximetry) on room air
4. Screening ECG QTc interval greater than 500ms by either a 12 lead or 6 lead ECG.
5. Concomitant drug-drug interactions (Artemether, Dapsone, Lumefantrine or Mefloquine amiodarone, digoxin, dofetilide, flecainide, procainamide, sotalol, or propafenone levofloxacin, ciprofloxacin, moxifloxacin, azithromycin, clarithromycin, erythromycin, ketoconazole, or itraconazole methadone sumatriptan, or zolmitriptan systemic chemotherapy.)
6. Already on active palliative care measures (Palliative performance score (PPS) less than 30%)
7. Hypersensitivity reaction to chloroquine, hydroxychloroquine or aminoquinolines
8. History of retinal disease due to previous use of 4-aminoquinoline
9. Prior documented and known at enrollment, retinal eye disease or maculopathy including but not limited to diabetic retinopathy, retinal detachment, retinitis pigmentosa or macular degeneration
10. Known glucose-6 phosphate dehydrogenase (G6PD) deficiency
11. Known Porphyria
12. Acute delirium
13. Inability to swallow oral study drug/placebo (even after crushed in the same manner as regular prescribed medications)
14. Diagnosis of immunodeficiency (e.g. HIV, transplantation) or receiving systemic steroid therapy (>10mg prednisone daily or equivalent) or any other form of immunosuppressive therapy prior to trial treatment
15. Women who are pregnant or breastfeeding

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-30 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of symptomatic fever >37.8, dry cough, or shortness of breath (resident/patient report or nurse observation) respiratory infection with confirmed PCR+ result for SARS-CoV-2. | baseline through day 90

SECONDARY OUTCOMES:
Requirement for admission to acute care hospital and/or ICU admission or death | baseline through day 90
Asymptomatic PCR+ SARS-CoV-2 test result | baseline, days 2, 5, 12, and 19
Time to clinical recovery (TTCR). | baseline through day 90

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Borrie, MB ChB, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou D, Dai SM, Tong Q. COVID-19: a recommendation to examine the effect of hydroxychloroquine in preventing infection and progression. J Antimicrob Chemother. 2020 Jul 1;75(7):1667-1670. doi: 10.1093/jac/dkaa114. PMID 32196083
- [Background] Borba MGS, Val FFA, Sampaio VS, Alexandre MAA, Melo GC, Brito M, Mourao MPG, Brito-Sousa JD, Baia-da-Silva D, Guerra MVF, Hajjar LA, Pinto RC, Balieiro AAS, Pacheco AGF, Santos JDO Jr, Naveca FG, Xavier MS, Siqueira AM, Schwarzbold A, Croda J, Nogueira ML, Romero GAS, Bassat Q, Fontes CJ, Albuquerque BC, Daniel-Ribeiro CT, Monteiro WM, Lacerda MVG; CloroCovid-19 Team. Effect of High vs Low Doses of Chloroquine Diphosphate as Adjunctive Therapy for Patients Hospitalized With Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Infection: A Randomized Clinical Trial. JAMA Netw Open. 2020 Apr 24;3(4):e208857. doi: 10.1001/jamanetworkopen.2020.8857. PMID 32330277
- [Background] Chen T, Wu D, Chen H, Yan W, Yang D, Chen G, Ma K, Xu D, Yu H, Wang H, Wang T, Guo W, Chen J, Ding C, Zhang X, Huang J, Han M, Li S, Luo X, Zhao J, Ning Q. Clinical characteristics of 113 deceased patients with coronavirus disease 2019: retrospective study. BMJ. 2020 Mar 26;368:m1091. doi: 10.1136/bmj.m1091. PMID 32217556
- [Background] Filatov A, Sharma P, Hindi F, Espinosa PS. Neurological Complications of Coronavirus Disease (COVID-19): Encephalopathy. Cureus. 2020 Mar 21;12(3):e7352. doi: 10.7759/cureus.7352. PMID 32328364
- [Background] Ghasemnejad-Berenji H, Ghaffari Novin M, Hajshafiha M, Nazarian H, Hashemi SM, Ilkhanizadeh B, Ghasemnejad T, Sadeghpour S, Ghasemnejad-Berenji M. Immunomodulatory effects of hydroxychloroquine on Th1/Th2 balance in women with repeated implantation failure. Biomed Pharmacother. 2018 Nov;107:1277-1285. doi: 10.1016/j.biopha.2018.08.027. Epub 2018 Aug 29. PMID 30257342
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Juurlink DN. Safety considerations with chloroquine, hydroxychloroquine and azithromycin in the management of SARS-CoV-2 infection. CMAJ. 2020 Apr 27;192(17):E450-E453. doi: 10.1503/cmaj.200528. Epub 2020 Apr 8. No abstract available. PMID 32269021
- [Background] Mao L, Jin H, Wang M, Hu Y, Chen S, He Q, Chang J, Hong C, Zhou Y, Wang D, Miao X, Li Y, Hu B. Neurologic Manifestations of Hospitalized Patients With Coronavirus Disease 2019 in Wuhan, China. JAMA Neurol. 2020 Jun 1;77(6):683-690. doi: 10.1001/jamaneurol.2020.1127. PMID 32275288
- [Background] McMichael TM, Currie DW, Clark S, Pogosjans S, Kay M, Schwartz NG, Lewis J, Baer A, Kawakami V, Lukoff MD, Ferro J, Brostrom-Smith C, Rea TD, Sayre MR, Riedo FX, Russell D, Hiatt B, Montgomery P, Rao AK, Chow EJ, Tobolowsky F, Hughes MJ, Bardossy AC, Oakley LP, Jacobs JR, Stone ND, Reddy SC, Jernigan JA, Honein MA, Clark TA, Duchin JS; Public Health-Seattle and King County, EvergreenHealth, and CDC COVID-19 Investigation Team. Epidemiology of Covid-19 in a Long-Term Care Facility in King County, Washington. N Engl J Med. 2020 May 21;382(21):2005-2011. doi: 10.1056/NEJMoa2005412. Epub 2020 Mar 27. PMID 32220208
- [Background] Troyer EA, Kohn JN, Hong S. Are we facing a crashing wave of neuropsychiatric sequelae of COVID-19? Neuropsychiatric symptoms and potential immunologic mechanisms. Brain Behav Immun. 2020 Jul;87:34-39. doi: 10.1016/j.bbi.2020.04.027. Epub 2020 Apr 13. PMID 32298803
- [Background] Verity R, Okell LC, Dorigatti I, Winskill P, Whittaker C, Imai N, Cuomo-Dannenburg G, Thompson H, Walker PGT, Fu H, Dighe A, Griffin JT, Baguelin M, Bhatia S, Boonyasiri A, Cori A, Cucunuba Z, FitzJohn R, Gaythorpe K, Green W, Hamlet A, Hinsley W, Laydon D, Nedjati-Gilani G, Riley S, van Elsland S, Volz E, Wang H, Wang Y, Xi X, Donnelly CA, Ghani AC, Ferguson NM. Estimates of the severity of coronavirus disease 2019: a model-based analysis. Lancet Infect Dis. 2020 Jun;20(6):669-677. doi: 10.1016/S1473-3099(20)30243-7. Epub 2020 Mar 30. PMID 32240634
- [Background] Albert DJ. Suppression of mouse killing by lateral hypothalamic infusion of atropine sulfate in the rat: a general behavioral suppression. Pharmacol Biochem Behav. 1980 May;12(5):681-4. doi: 10.1016/0091-3057(80)90148-3. PMID 7190303